CLINICAL TRIAL: NCT01935297
Title: Safety, Applicability and Outcome of Regular Exercise Training After Transcatheter Aortic Valve Implantation
Brief Title: Exercise Training After Transcatheter Aortic Valve Implantation
Acronym: SPORT:TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Deutsches Herzzentrum Muenchen (Other); Klinikum der Universitaet Muenchen, Grosshadern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F/14/12
Record Dates: First submitted 2013-07-05; First posted 2013-09-05 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Transcatheter Aortic Valve Replacement
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Active Comparator): 8 weeks of supervised, structured, combined endurance and resistance training
  Interventions: Behavioral: Exercise
- Control (No Intervention): Patients receive usual care, regular exercise is not recommended but also not prohibited

INTERVENTIONS:
Behavioral: Exercise — endurance and resistance exercise 3x/week for 8 weeks
  Arms: Exercise

SUMMARY:
This pilot study will evaluate the effect of a rehabilitative exercise training on exercise capacity in patients after percutaneous aortic valve replacement. It will additionally evaluate the safety of such an approach and the effect on life quality. We hypothesize that regular structured exercise improves exercise capacity in these patients beyond the sole effect of the valve procedure.

DETAILED DESCRIPTION:
The study will include 30 patients and randomize them in a 1:1-fashion to either a training or a usual care group. The training group will undergo 8 weeks of combined endurance and resistance training according to a standard protocol, but with individual adjustment if required. The usual care group will receive general advice but no structured exercise program. Exercise capacity is assessed by cardiopulmonary exercise testing and by the 6 minute walk test prior to and after the intervention period. In addition, life quality will be assessed by validated questionnaires, while safety will be assessed by recording adverse events and by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

patients up to 6 months after transcatheter aortic valve implantation

Exclusion Criteria:

inability to perform exercise on bicycles valve dysfunction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change of peak oxygen uptake | Baseline to 8 weeks

SECONDARY OUTCOMES:
Change of quality of life | Baseline to 8 weeks
  Assessed by SF-12 and KCCQ questionnaires

OTHER OUTCOMES:
Change of valve function | Baseline to 8 weeks
  Assessed by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Axel Pressler, MD, Principal Investigator — Prevention, Rehabilitation & Sports Medicine, Technische Universität München, Germany
Locations (1):
- Department of prevention, rehabilitation and sports medicine, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Pressler A, Forschner L, Hummel J, Haller B, Christle JW, Halle M. Long-term effect of exercise training in patients after transcatheter aortic valve implantation: Follow-up of the SPORT:TAVI randomised pilot study. Eur J Prev Cardiol. 2018 May;25(8):794-801. doi: 10.1177/2047487318765233. Epub 2018 Mar 19. PMID 29553289
- [Derived] Pressler A, Christle JW, Lechner B, Grabs V, Haller B, Hettich I, Jochheim D, Mehilli J, Lange R, Bleiziffer S, Halle M. Exercise training improves exercise capacity and quality of life after transcatheter aortic valve implantation: A randomized pilot trial. Am Heart J. 2016 Dec;182:44-53. doi: 10.1016/j.ahj.2016.08.007. Epub 2016 Aug 26. PMID 27914499